CLINICAL TRIAL: NCT06435650
Title: The Use of Mindful Compassion and Cannabis Suppositories for Anal Pain Among Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Metropolitan University (Other)
Responsible Party: Principal Investigator, Samantha Banbury, Principal Investigator, London Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: London Metropolitan University
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Pain;Sexual Intercourse;M
Keywords: Mindful-compassion; Well-being; Sexual self efficacy; Sexual functioning

STUDY DESIGN:
Intervention Model Description: The study phase is not applicable as whilst cannabis suppositories are part of this research study, participants are not randomised into cannabis groups. Participants would already be using cannabis suppositories for at least one month and are used as part of sexual intimacy.
  Randomisation was based on whether participants were using cannabis suppositories and consisted of one of four groups, including a cannabis suppository-only group, mindful- compassion only group, a combined mindful-compassion and cannabis suppository group and a care-as-usual group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful-compassion group (Experimental): Online mindful-compassion weekly for four weeks
  Interventions: Behavioral: Mindful-compassion
- Mindful-compassion and Cannabis suppository (Experimental): Participants were not prescribed cannabis as part of this study. Participants had been for at least one month before participating in the study. Participants used cannabis suppositories each time they engaged in anal intercourse (recipient). The average dose, based on participant reports, was approximately 500mg.
  Online mindful-compassion weekly for four weeks
  Interventions: Combination Product: Cannabis suppositories and mindful-compassion for anal pain

INTERVENTIONS:
Combination Product: Cannabis suppositories and mindful-compassion for anal pain — This is a combined intervention that includes mindful-compassion and cannabis suppositories for anal pain
  Arms: Mindful-compassion and Cannabis suppository
Behavioral: Mindful-compassion — Mindful-compassion
  Arms: Mindful-compassion group

SUMMARY:
Research aim: To determine how an online mindful-compassion intervention adjunct with cannabis suppositories might reduce anal pain during sexual intimacy among men who have sex with men. Outcomes are also hoped to increase sexual functioning, well-being and sexual self-efficacy.

Research intention: If the combined mindful compassion and cannabis suppository intervention reduces anal pain and supports sexual and general well-being, then this research would be repeated on a larger scale targeting psychosexual services.

A brief overview of the intervention:

Anal pain is pain experienced in the anus during anal penetration with a penis or other objects. Most research on anal pain during sexual intimacy has centred on men who have sex with men. Mindfulness has been anecdotally discussed in reducing symptoms of anal pain in men who have sex with men. A novel approach to pain management includes medical cannabis, which can be cannabidiol, tetrahydrocannabinol or both. Anal suppositories do not create a euphoric high in the same way as oral use, including inhalation.

Quantitatively, randomisation will be based on whether participants use cannabis suppositories or not. This study does not randomise to cannabis groups owing to the legalities in the United Kingdom. Participants included fifty-two consenting participants. Of these, thirty-three were using cannabis suppositories. The intervention was delivered for one month, and the follow-up was at twelve weeks. Qualitatively, participants were asked approximately eight open-ended feedback questions throughout the study.

DETAILED DESCRIPTION:
Research looking at mindfulness-based interventions or the use of medical cannabis to support sexual pain is limited, and often, sexual pain goes unreported, which might lead to compromised psychological well-being. Additionally, sexual problems associated with pain and related emotional suffering are frequently overlooked in patients with sexual pain. This research aims to establish the effectiveness of an online mindful compassion intervention adjunct with cannabis suppositories to help minimise sexual pain and increase well-being. This research decided to deliver mindful compassion online because it would economically target a more comprehensive and diverse group. This preliminary study examined how a mindful compassion intervention combined with cannabis suppositories might help minimise sexual pain whilst improving sexual function, well-being, and sexual self-efficacy.

The main exercises included mindfulness, breathing, relaxation techniques, Mindfulness of the senses and body, and understanding the self. These exercises incorporated the three-model system of emotions, how to attend to the cognitive and physical patterns associated with painful sex, and towards acceptance and self-compassion with fewer symptoms. The mindful-compassion intervention included psychosexual education and anal pain, the three-model system of emotions and sexual pain, practising mindful compassion and graded practice and self-care, efficacy, and the relationship with anatomy.

Homework exercises, including education, training, modelling, and enablement, were encouraged. Feedback and support, along with discussing the educational components, training, modelling, and enablement, were addressed throughout this study.

The development of mindful compassion intervention has been based on a taxonomy of behavioural change techniques. This has been used because the taxonomy of behavioural change techniques has been rigorously tested to evidence the effectiveness in supporting interventions associated with change behaviour. The 93 behaviour change techniques are the active ingredients of behaviour change, and each intervention is likely to consist of more than one behaviour change technique and serve as having more than one function. The intervention in this study included twelve domains, of which twenty-three out of the 93 behaviour change techniques listed in the behavioural change technique taxonomy were identified. The selection of these domains used a triangulation process to ensure consistency in mapping the behaviour change techniques to the intervention.

Randomisation was based on whether participants were already using cannabis suppositories or not. Those who did use cannabis suppositories as part of their sex life would have been doing so for at least a month. There was a total of four groups, including a cannabis suppository-only group, a mindful-compassion-only group, a combined mindful compassion and cannabis suppository group and a care-as-usual group.

ELIGIBILITY:
Inclusion Criteria:

* Participants were allocated to cannabis only, and cannabis adjunct groups would already be using cannabis suppositories.
* Must have engaged in anal sex within the last month
* Must be based in the United Kingdom
* Must have experienced anal sexual pain
* An absence of co-occurring difficulties
* Must be aged 18 years or older
* Must be able to read and write English.
* Patient health screening score must range between 0-9 mild
* Generalised anxiety disorder screening score must range between 0-9, mild

Exclusion Criteria:

* Have not attempted anal intercourse in the last month
* Have co-occurring difficulties
* Aged below 18 years old
* Reading and writing English difficulties
* Not experiencing anal pain during sexual intercourse.
* Patient health screening score ranged between moderate to severe - 10-27
* Generalised anxiety screening score ranged between 10- 21.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who have sex with men Those who identify as male
Enrollment: 52 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Changes in levels of anal pain taken at weeks 0, 4 and 12 | 0, 4 and 12 weeks
  The frequency and severity of pain during anal sex, this is a 5-point Likert-type scale which ranges from never (5) to all the time (1) and no anal pain (5) to severe anal pain (1). The Cronbach alpha in this study= 0.70.
Changes in sexual functioning taken at weeks 0, 4 and 12 | 0, 4 and 12 weeks
  This is an 11-item questionnaire which focuses on sexual functioning including sexual desire, arousal and satisfaction and erectile functioning. The response categories include 0= not at all to 5= always or 0= no problem to 5= big problem (this varied pending question). The Cronbach alpha in this study = 0.75.
Changes in levels of well-being at weeks 0,4 and 12 | 0, 4 and 12 weeks
  This is a 7-item questionnaire with 5 response categories looking at functioning and feeling aspects of well-being. The response categories include 1=none of the time to 5=all of the time. Cronbach alpha- 0.89-0.91. There is no reverse scoring. Scores range from 7 to 35 where the latter is the highest level of wellbeing. The Cronbach alpha in this study = 0.85.
Changes in levels of sexual self-efficacy at weeks 0, 4 and 12 | 0, 4 and 12 weeks
  This is a 10-item questionnaire which focuses on sexual confidence and behaviour. The response categories include: 1 is the lowest level of self-efficacy and 10 is the highest. There are no reverse questions. Cronbach's alpha is α =0.88 (high). This questionnaire has been adapted to reflect the participants in a study looking at sexual self-efficacy and sexual function. Less than 5% of the original questionnaire remains. The Cronbach alpha in this study= 0.83.
Changes in levels of mindful-compassion | 0, 4 and 12
  This is a 12-item measure with 5 response categories, 1 = almost never to 5 = almost always, with higher scores indicating higher levels of self-compassion. The questionnaire measures self-kindness vs. self-judgement, common humanity vs. isolation, and mindfulness vs. over-identification with painful thoughts and emotions. Reliability Cronbach's alphas range between 0.68 and 0.78. The Cronbach alpha in this study was 0.73.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Banbury, Principal Investigator — London Metropolitan University
Locations (1):
- Samantha Banbury, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barach E, Slavin MN, Earleywine M. Cannabis and Vulvodynia Symptoms: A Preliminary Report. Cannabis. 2020 Jul 3;3(2):139-147. doi: 10.26828/cannabis.2020.02.001. PMID 33426502
- [Result] Bloomfield MA, Ashok AH, Volkow ND, Howes OD. The effects of Delta9-tetrahydrocannabinol on the dopamine system. Nature. 2016 Nov 17;539(7629):369-377. doi: 10.1038/nature20153. PMID 27853201
- [Result] Boardman LA, Stockdale CK. Sexual pain. Clin Obstet Gynecol. 2009 Dec;52(4):682-90. doi: 10.1097/GRF.0b013e3181bf4a7e. PMID 20393420
- [Result] Brenneisen R, Egli A, Elsohly MA, Henn V, Spiess Y. The effect of orally and rectally administered delta 9-tetrahydrocannabinol on spasticity: a pilot study with 2 patients. Int J Clin Pharmacol Ther. 1996 Oct;34(10):446-52. PMID 8897084
- [Result] Brotto LA, Bergeron S, Zdaniuk B, Driscoll M, Grabovac A, Sadownik LA, Smith KB, Basson R. A Comparison of Mindfulness-Based Cognitive Therapy Vs Cognitive Behavioral Therapy for the Treatment of Provoked Vestibulodynia in a Hospital Clinic Setting. J Sex Med. 2019 Jun;16(6):909-923. doi: 10.1016/j.jsxm.2019.04.002. Epub 2019 May 15. PMID 31103481
- [Result] Carey RN, Connell LE, Johnston M, Rothman AJ, de Bruin M, Kelly MP, Michie S. Behavior Change Techniques and Their Mechanisms of Action: A Synthesis of Links Described in Published Intervention Literature. Ann Behav Med. 2019 Jul 17;53(8):693-707. doi: 10.1093/abm/kay078. PMID 30304386
- [Result] ElSohly MA, Gul W, Walker LA. Pharmacokinetics and Tolerability of Delta9-THC-Hemisuccinate in a Suppository Formulation as an Alternative to Capsules for the Systemic Delivery of Delta9-THC. Med Cannabis Cannabinoids. 2018 Jun 12;1(1):44-53. doi: 10.1159/000489037. eCollection 2018 Jun. PMID 34676321
- [Result] Fisher E, Moore RA, Fogarty AE, Finn DP, Finnerup NB, Gilron I, Haroutounian S, Krane E, Rice ASC, Rowbotham M, Wallace M, Eccleston C. Cannabinoids, cannabis, and cannabis-based medicine for pain management: a systematic review of randomised controlled trials. Pain. 2021 Jul 1;162(Suppl 1):S45-S66. doi: 10.1097/j.pain.0000000000001929. PMID 32804836
- [Result] Kondrad E. Medical marijuana for chronic pain. N C Med J. 2013 May-Jun;74(3):210-1. No abstract available. PMID 23940889
- [Result] Liang AL, Gingher EL, Coleman JS. Medical Cannabis for Gynecologic Pain Conditions: A Systematic Review. Obstet Gynecol. 2022 Feb 1;139(2):287-296. doi: 10.1097/AOG.0000000000004656. PMID 35104069
- [Result] Libman E, Rothenberg I, Fichten CS, Amsel R. The SSES-E: a measure of sexual self-efficacy in erectile functioning. J Sex Marital Ther. 1985 Winter;11(4):233-47. doi: 10.1080/00926238508405450. PMID 4078907
- [Result] Vaishnava PP, Kimball CW, Matykiewicz JL, Fradin FY, Shenoy GK, Montano PA. Extended x-ray-absorption fine-structure observation of collinear ordering of Fe-Sn-Fe atoms in the Chevrel-phase superconductor SnFe0.05Mo6S8. Phys Rev B Condens Matter. 1986 Oct 1;34(7):4599-4603. doi: 10.1103/physrevb.34.4599. No abstract available. PMID 9940251
- [Result] Haug T. Tolerance to the depressant effects of diazepam in the drug discrimination paradigm. Pharmacol Biochem Behav. 1984 Sep;21(3):409-15. doi: 10.1016/s0091-3057(84)80103-3. PMID 6494210
- [Result] Nercessian TR, Banbury S, Chandler C. A Systematic Review Looking at Anodyspareunia Among Cisgender Men and Women. J Sex Marital Ther. 2023;49(7):829-841. doi: 10.1080/0092623X.2023.2196265. Epub 2023 Apr 23. PMID 37089031
- [Result] Suarez Guglielmini H, Schurmann Ruppert R, O'Ryan Costa P. [Measles. Clinical and anatomo-pathologic study]. Rev Chil Pediatr. 1966 Aug-Sep;37(8):477-84. No abstract available. Spanish. PMID 5986896
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Rycroft-Malone J, Gradinger F, Griffiths HO, Crane R, Gibson A, Mercer S, Anderson R, Kuyken W. Accessibility and implementation in the UK NHS services of an effective depression relapse prevention programme: learning from mindfulness-based cognitive therapy through a mixed-methods study. Southampton (UK): NIHR Journals Library; 2017 Mar. Available from http://www.ncbi.nlm.nih.gov/books/NBK425272/ PMID 28368561
- [Result] Bowman BH, Barnett DR, Hodgkinson KT, Schneider RG. Chemical characterization of haemoglobin G-St-I. Nature. 1966 Sep 17;211(5055):1305-6. doi: 10.1038/2111305a0. No abstract available. PMID 5969816
- [Result] Munoz M, Munoz A, Gonzalez A. Distribution, morphology, and central projections of mesencephalic trigeminal neurons in the frog Rana ridibunda. Anat Rec. 1993 Jan;235(1):165-77. doi: 10.1002/ar.1092350117. PMID 8417625
- [Result] Smith EJ, Palevsky S. Salt poisoning in a two-year-old child. Am J Emerg Med. 1990 Nov;8(6):571-2. doi: 10.1016/0735-6757(90)90183-z. No abstract available. PMID 2222612
- [Result] Antonelli AR, Bellotto R, Bertazzoli M, Busnelli GP, Nunez Castro M, Felisati G, Romagnoli M. Auditory brain stem response test battery for multiple sclerosis patients: evaluation of test findings and assessment of diagnostic criteria. Audiology. 1986;25(4-5):227-38. PMID 3566631